CLINICAL TRIAL: NCT04623437
Title: Comprehensive Antineoplastic Therapy Adverse Events Monitoring and Report
Brief Title: Responsible Side Effects Management in Oncology
Acronym: R-SEMO
Status: Completed | Type: Observational
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Robert Šeparović, PhD MD, University Hospital Sestre Milosrdnice
Other Study IDs: 2312201522122016
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Pharmacovigilance; Oncology; Antineoplastic Treatment
Keywords: pharmacovigilance in oncology; antineoplastic treatment; adverse events
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of pharmacovigilance in oncology. Monitoring and management of AEs during antineoplastic treatment.

DETAILED DESCRIPTION:
Monitoring and management of AE's during antineoplastic treatment. Comparison of AE's reported by patient with the ones recognised by the oncologist, and vice versa, during antineoplastic treatment.

ELIGIBILITY:
Inclusion Criteria:

all cancer patients receiving systemic antineoplastic treatment, ECOG 0-2

Exclusion Criteria:

age <18, >75; other active and severe comorbidities; no solid cancer; IUC patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all cancer patients actively receiving systemic antineoplastic treatment, ECOG 0-2
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
comparison of perspectives | may 2016 until october 2016
  comparison between patient's and oncologist's perspective on severity of AE's during antineoplastic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UHC Sestre milorsdnice, Zagreb, Croatia, Europe, Croatia